CLINICAL TRIAL: NCT00398281
Title: Detection of Prostate Cancer With Contrast-Enhanced Ultrasound After Treatment With Dutasteride
Brief Title: Dutasteride Followed By Ultrasound-Guided Biopsy in Finding Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ethan J. Halpern, Kimmel Cancer Center at Thomas Jefferson University - Philadelphia
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Diagnostic
Other Study IDs: CDR0000513051; TJUH-06F-145; NCT00330057 (obsolete NCT alias)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

ARMS (2):
- Arm I (Experimental): Patients receive oral dutasteride once daily on days 1-14.
  Interventions: Drug: dutasteride
- Arm II (Placebo Comparator): Patients receive oral placebo once daily on days 1-14.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: dutasteride — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Diagnostic procedures, such as ultrasound-guided biopsy, may help find prostate cancer. Dutasteride may improve the ability of ultrasound-guided biopsy to find prostate cancer. It is not yet known whether dutasteride followed by ultrasound-guided biopsy is more effective than a placebo followed by ultrasound-guided biopsy in finding prostate cancer.

PURPOSE: This randomized phase III trial is studying dutasteride and ultrasound-guided biopsy to see how well they find prostate cancer compared with a placebo and ultrasound-guided biopsy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of dutasteride followed by contrast-enhanced, ultrasound-guided targeted biopsy in detecting prostate cancer.
* Determine the detection rate of prostate cancer with targeted biopsy using contrast-enhanced ultrasound combined with dutasteride.
* Determine the efficacy of targeted biopsy using contrast-enhanced ultrasound vs systematic biopsy in diagnosing clinically significant prostate cancer.
* Determine the reduction in post-biopsy bleeding after dutasteride in these patients.
* Determine the cost effectiveness of this regimen in these patients.

OUTLINE: This is a prospective, double-blind, placebo-controlled, randomized study. Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral dutasteride once daily on days 1-14.
* Arm II: Patients receive oral placebo once daily on days 1-14. On day 14, patients in both arms undergo blood collection and contrast-enhanced (perflutren protein-type A microspheres) transrectal ultrasound. Conventional gray-scale imaging, color Doppler imaging, and power Doppler imaging are performed. Biopsies are then performed; first up to 6 targeted ultrasound-guided biopsies and then up to 12 systematic biopsies.

After completion of study procedures, patients are followed at 1 day.

PROJECTED ACCRUAL: A total of 450 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Suspected prostate cancer due to 1 of the following criteria:

  * Prior abnormal digital rectal exam
  * Elevated prostate-specific antigen (PSA) ≥ 2.6 ng/mL within the past 90 days
  * PSA velocity > 0.75 ng/mL/year
* Must be planning to undergo a transrectal ultrasound with biopsy

PATIENT CHARACTERISTICS:

* Must be in adequate physical health to tolerate a prolonged transrectal examination and biopsy
* Must not be clinically unstable, severely ill, or moribund

PRIOR CONCURRENT THERAPY:

* More than 30 days since prior biopsy of the prostate
* More than 1 week since prior acetylsalicylic acid or blood thinner
* More than 30 days since prior participation in a clinical trial involving an investigational drug
* No prior therapy for prostate cancer
* No other concurrent 5-alpha reductase inhibitor

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of short-term dutasteride in improving prostate cancer detection
Detection rate of prostate cancer
Cost effectiveness of contrast-enhanced ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ethan J. Halpern, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Halpern EJ, Gomella LG, Forsberg F, McCue PA, Trabulsi EJ. Contrast enhanced transrectal ultrasound for the detection of prostate cancer: a randomized, double-blind trial of dutasteride pretreatment. J Urol. 2012 Nov;188(5):1739-45. doi: 10.1016/j.juro.2012.07.021. Epub 2012 Sep 19. PMID 22998915